CLINICAL TRIAL: NCT04337112
Title: The Expanded Access Use of Viltolarsen for the Treatment of Duchenne Muscular Dystrophy (DMD) Amenable to Exon 53 Skipping
Brief Title: The Expanded Access Use of Viltolarsen in Duchenne Muscular Dystrophy With Confirmed Exon 53 Amenable Mutation
Status: Approved for marketing | Type: Expanded Access
Sponsor: NS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VILT-501
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Muscular Dystrophy, Duchenne; DMD
Keywords: Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Muscular Disorders, Atrophic; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases; Genetic Diseases, Inborn; Genetic Diseases, X-Linked | interventions — viltolarsen

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: viltolarsen — Intravenous (IV) infusions, weekly, at 80mg/kg, once weekly (approximately every 7 days).
  Other Names: NS-065/NCNP-01

SUMMARY:
This is an open label expanded access program for boys, 3 to 12 years old, for the treatment of Duchenne muscular dystrophy (DMD) with confirmed mutation(s) in the dystrophin gene that is amenable to skipping of exon 53.

DETAILED DESCRIPTION:
This expanded access program is designed to provide access to viltolarsen in patients with DMD with confirmed mutation(s) in the dystrophin gene amenable to skipping of exon 53, who in the opinion and clinical judgement of the treating physician, would benefit from treatment with viltolarsen.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 3 and ≤ 12 years of age
* Clinical signs compatible with DMD
* Confirmed DMD mutation(s) in the dystrophin gene that is amenable to skipping of exon 53 to restore the dystrophin messenger ribonucleic acid (mRNA) reading frame
* Able to walk independently without assistive device
* Not able to participate in a Phase 3 trial

Exclusion Criteria:

* Chronic systemic fungal or viral infections
* An acute illness within 4 weeks prior to the first dose of viltolarsen
* Symptomatic cardiomyopathy
* Patient has a previous or ongoing medical condition, medical history, physical findings, or laboratory abnormality that could affect participant safety in the opinion of the treating physician
* Surgery within the 3 months prior to the first anticipated administration of viltolarsen and in the opinion of the treating physician would impact weekly treatment schedule
* Positive test results for hepatitis B antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) antibody at screening
* Currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to the first dose of viltolarsen
* Previously enrollment in any viltolarsen study.
* Currently taking any other exon skipping agent or has taken any other exon skipping agent within 2 weeks prior to the first dose of viltolarsen (would need to be discontinued in order to be eligible)
* Any gene therapy for DMD
* Inadequate renal function as defined by a serum cystatin C > 1.5 x upper limit of normal (ULN). If the value is > 1.5 x ULN then the measurement can be repeated once. If repeat measurement is still > 1.5 x ULN then the patient should be excluded.

Ages: 3 Years to 12 Years | Sex: Male
Age Groups: Child